CLINICAL TRIAL: NCT01976091
Title: Phase I/IIA Gene Transfer Clinical Trial for LGMD2D (Alpha-Sarcoglycan Deficiency) Using scAAVrh74.tMCK.hSGCA
Brief Title: A Gene Transfer Therapy Study to Evaluate the Safety of SRP-9004 (Patidistrogene Bexoparvovec) in Participants With Limb-Girdle Muscular Dystrophy, Type 2D (LGMD2D)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9004-101; 5U01AR060911 (NIH)
Record Dates: First submitted 2013-07-24; First posted 2013-11-05 (Estimated); Results first posted 2022-04-01 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-04

CONDITIONS: Limb-Girdle Muscular Dystrophy, Type 2D
Keywords: limb girdle muscular dystrophy; LGMD2D; alpha-sarcoglycan; gene transfer; adeno-associated virus
MeSH Terms: conditions — Sarcoglycanopathies; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1A: SRP-9004 Low Dose (Single Limb Perfusion) (Experimental): Non-ambulant participants with LGMD2D will receive 1 low dose of SRP-9004 via ILI to a single limb on Day 0.
  Interventions: Genetic: SRP-9004
- Cohort 1B Low Dose (Bilateral Limb Perfusion) (Experimental): Participants with LGMD2D will receive 1 low dose of SRP-9004 via ILI to both limbs on Day 0.
  Interventions: Genetic: SRP-9004
- Cohort 2 High Dose (Bilateral Limb Perfusion) (Experimental): Participants with LGMD2D will receive 1 high dose of SRP-9004 via ILI to both limbs on Day 0.
  Interventions: Genetic: SRP-9004

INTERVENTIONS:
Genetic: SRP-9004 — Isolated Limb Infusion (ILI)
  Other Names: patidistrogene bexoparvovec

SUMMARY:
This is an open-label, dose escalation gene transfer therapy study evaluating the safety of SRP-9004 (patidistrogene bexoparvovec) via isolated limb infusion (ILI) administration in approximately 6 participants with LGMD2D.

ELIGIBILITY:
Key Inclusion Criteria:

* Cohort 1A must be adult and wheelchair-dependent; Cohorts 1B and 2 will be participants of age 7 or older.
* Confirmed alpha-sarcoglycan deficiency or identified sarcoglycan alpha (SGCA) deoxyribonucleic acid (DNA) mutation.
* Participants enrolled in Cohorts 1B or 2 must be able to walk independently, but must exhibit signs of lower extremity weakness (that is, a Gowers' sign, use a handrail for climbing stairs) and walk ≤80% of predicted distance on the 6 minute walk test (6MWT) based on normative data.

Key Exclusion Criteria:

* Active viral infection based on clinical observations.
* The presence of SGCA mutations without weakness or loss of function.
* Symptoms or signs of cardiomyopathy.
* Serological evidence of human immunodeficiency virus (HIV), Hepatitis B, or C infection.
* Diagnosis of (or ongoing treatment for) an autoimmune disease.
* Participants with AAVrh74 or AAV8 binding antibody titers ≥ 1:50 as determined by enzyme-linked immunosorbent assay (ELISA) immunoassay.

Other inclusion/exclusion criteria apply.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.

REFERENCES:
- [Background] Mendell JR, Chicoine LG, Al-Zaidy SA, Sahenk Z, Lehman K, Lowes L, Miller N, Alfano L, Galliers B, Lewis S, Murrey D, Peterson E, Griffin DA, Church K, Cheatham S, Cheatham J, Hogan MJ, Rodino-Klapac LR. Gene Delivery for Limb-Girdle Muscular Dystrophy Type 2D by Isolated Limb Infusion. Hum Gene Ther. 2019 Jul;30(7):794-801. doi: 10.1089/hum.2019.006. Epub 2019 Apr 19. PMID 30838895
- [Background] Mendell JR, Rodino-Klapac LR, Rosales XQ, Coley BD, Galloway G, Lewis S, Malik V, Shilling C, Byrne BJ, Conlon T, Campbell KJ, Bremer WG, Taylor LE, Flanigan KM, Gastier-Foster JM, Astbury C, Kota J, Sahenk Z, Walker CM, Clark KR. Sustained alpha-sarcoglycan gene expression after gene transfer in limb-girdle muscular dystrophy, type 2D. Ann Neurol. 2010 Nov;68(5):629-38. doi: 10.1002/ana.22251. PMID 21031578
- [Background] Mendell JR, Rodino-Klapac LR, Rosales-Quintero X, Kota J, Coley BD, Galloway G, Craenen JM, Lewis S, Malik V, Shilling C, Byrne BJ, Conlon T, Campbell KJ, Bremer WG, Viollet L, Walker CM, Sahenk Z, Clark KR. Limb-girdle muscular dystrophy type 2D gene therapy restores alpha-sarcoglycan and associated proteins. Ann Neurol. 2009 Sep;66(3):290-7. doi: 10.1002/ana.21732. PMID 19798725

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with limb-girdle muscular dystrophy, type 2D (LGMD2D) were enrolled into 3 cohorts: Cohort 1A (non-ambulant adult participants), Cohort 1B (pediatric participants), and Cohort 2 (pediatric participants).
Groups:
- Cohort 1A: SRP-9004: SRP-9004 was administered once by Isolated Limb Infusion (ILI) to a single limb on Day 0. The administered dose was 1*10^12 vector genomes per kilogram body weight (vg/kg). Dose determined via supercoiled titer method.
- Cohort 1B: SRP-9004: SRP-9004 was administered once by ILI to both limbs on Day 0. The participants received a total dose of 2*10^12 vg/kg split between the two extremities (1*10^12 vg/kg per limb). Dose determined via supercoiled titer method.
- Cohort 2: SRP-9004: SRP-9004 was administered once by ILI to both limbs on Day 0. The participants received a total dose of 6*10^12 vg/kg split between the two extremities (3*10^12 vg/kg per limb). Dose determined via supercoiled titer method.
Period: Overall Study
Arm/Group | Cohort 1A: SRP-9004 | Cohort 1B: SRP-9004 | Cohort 2: SRP-9004
Started | 1 | 3 | 2
Received at Least 1 Dose of Study Drug | 1 | 3 | 2
Completed | 1 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received at least 1 administration of SRP-9004 during the study.
Groups:
- Cohort 1A: SRP-9004: SRP-9004 was administered once by ILI to a single limb on Day 0. The administered dose was 1*10^12 vector genomes per kilogram body weight (vg/kg). Dose determined via supercoiled titer method.
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: SRP-9004 | Cohort 1B: SRP-9004 | Cohort 2: SRP-9004 | Total
Number analyzed (Participants) | 1 | 3 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (NA) — Only 1 participant was enrolled into Cohort 1A. Therefore, the Standard Deviation (SD) is not applicable to this arm. | 10 (2.65) | 10 (2.83) | 16.5 (16.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 0 | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 3 | 2 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs).
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered study drug related. An AE was considered serious if, in the view of the investigator or sponsor, it resulted in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Treatment-related Treatment Emergent Adverse Event (TEAE) is defined as an TEAE that was classified by the investigator as related to treatment.
Time Frame: Up to 2 Years
Population: The FAS included all participants who received at least 1 administration of SRP-9004.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: SRP-9004 | Cohort 1B: SRP-9004 | Cohort 2: SRP-9004
Number analyzed (Participants) | 1 | 3 | 2
Participants
  Adverse Events | 1 | 3 | 2
  Serious Adverse Events | 0 | 2 | 1
  Treatment Related TEAEs | 1 | 3 | 2

2. Secondary Outcome: Change From Baseline of the Distance Walked in 6 Minutes (6MWT)
Description: The 6MWT was performed by standardized procedures for all participants. Participants were asked to walk a set course in 6 minutes (timed), and the distance walked (in meters) was recorded.
Time Frame: Baseline, Up to 2 Years
Population: The FAS included all participants who received at least 1 administration of SRP-9004. Here, Overall "Number of Participants Analyzed" signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Cohort 1A: SRP-9004 | Cohort 1B: SRP-9004 | Cohort 2: SRP-9004
Number analyzed (Participants) | 1 | 2 | 1
Meters | NA (NA) — Only 1 participant was enrolled into Cohort 1A. The participant was non-ambulatory at baseline and was not able to complete the 6MWT. Therefore, the Mean and SD are not applicable to this arm. | -66.0 (77.78) | 29.0 (NA) — Only 1 participant had evaluable data in this arm. Therefore, the SD is not applicable to this arm.

ADVERSE EVENTS:
Time Frame: Baseline up to 2 Years
Description: The FAS included all participants who were enrolled and received at least 1 dose of SRP-9004 during the study.
Arm/Group | Cohort 1A: SRP-9004 | Cohort 1B: SRP-9004 | Cohort 2: SRP-9004
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/3 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A: SRP-9004 (N=1) | Cohort 1B: SRP-9004 (N=3) | Cohort 2: SRP-9004 (N=2)
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myoglobinuria (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A: SRP-9004 (N=1) | Cohort 1B: SRP-9004 (N=3) | Cohort 2: SRP-9004 (N=2)
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 2
Viral infection (Infections and infestations) | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Adrenal suppression (Endocrine disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Myoglobinuria (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT01976091/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT01976091/SAP_001.pdf